CLINICAL TRIAL: NCT05191953
Title: Erector Spinae Plane Block Versus Its Combination With Superficial Parasternal Intercostal Plane Block for Postoperative Pain After Cardiac Surgery: A Prospective, Randomized, Double-blind Study
Brief Title: ESPB vs.Combination of ESPB and Superficial PIPB in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ESPBPIPB0255
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia; Analgesia; Acute Pain; Patient Controlled Analgesia
Keywords: Regional Anesthesia; Acute Pain Scores; Morphine Consumption
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used for the purpose of assigning each patient. A researcher not involved in patient followup will use the web based "Research Randomizer'' (Urbaniak and Plous 2013) tool in order to assign each participation number into a random group with a 1:1 ratio.
  A nurse that is not an active investigator in the study will have each participant choose an envelope that contains the study participation number. An assistant not active in the study will inform the anesthetist who will administer the block/blocks about which group the patient is in, immediately prior to administration. Researchers, patients, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB (Active Comparator): A bilateral ESPB (40 ml, %0.25 bupivacaine, totally) + IV morphine-PCA
  Interventions: Procedure: Bilateral ultrasound-guided ESPB
- Group ESPB+Superficial PIPB (Active Comparator): A bilateral ESPB (40 ml, %0.25 bupivacaine, totally) and a bilateral superficial PIPB (20 ml, %0.25 bupivacaine, totally) + IV morphine-PCA
  Interventions: Procedure: Bilateral ultrasound-guided ESPB and superficial PIPB

INTERVENTIONS:
Procedure: Bilateral ultrasound-guided ESPB — Bilateral ultrasound-guided ESPB (total of 40 ml, 0.25% bupivacaine) will be performed.
  Intraoperative analgesia:
  At the end of the surgery, all patients will be given 0.05 mg/kg morphine IV. Postoperative analgesia: Paracetamol 1 gr IV (every 6 hours) and IV PCA of 0.5 mg/ml morphine (demand dose 20μg/kg; lock out interval 6-10 min.; the 4-hour limit will be 80% of the total calculated dose). In cases where rescue analgesia is required (NRS score ≥4) tramadol 100 mg IV will be infused within 30 minutes (max. 300 mg / day). For postoperative nausea and vomiting prophylaxis, patients will be routinely administered ondansetron 4 mg IV 20 minutes before extubation, in the intensive care unit.
  Arms: Group ESPB
Procedure: Bilateral ultrasound-guided ESPB and superficial PIPB — Bilateral ultrasound-guided ESPB (total of 40 ml, %0.25 bupivacaine) and Superficial PIPB (total of 20 ml, %0.25 bupivacaine) will be performed.
  Intraoperative analgesia:
  At the end of the surgery, all patients will be given 0.05 mg/kg morphine IV. Postoperative analgesia: Paracetamol 1 gr IV (every 6 hours) and IV PCA of 0.5 mg/ml morphine (demand dose 20μg/kg; lock out interval 6-10 min.; the 4-hour limit will be 80% of the total calculated dose). In cases where rescue analgesia is required (NRS score ≥4) tramadol 100 mg IV will be infused within 30 minutes (max. 300 mg / day). For postoperative nausea and vomiting prophylaxis, patients will be routinely administered ondansetron 4 mg IV 20 minutes before extubation, in the intensive care unit.
  Arms: Group ESPB+Superficial PIPB

SUMMARY:
Cardiac surgery is associated with significant postoperative pain. Pain control is an essential part of enhanced recovery protocols. The aim of this study is to evaluate and compare the analgesic efficacies of erector spinae plane block (ESPB) and the combination of ESPB and superficial parasternal intercostal plane block (PIPB) in patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Many regional techniques have been used to manage postoperative pain in cardiac surgery, including thoracic epidural anesthesia, paravertebral, intercostal nerve block, intrathecal spinal morphine, and local infiltration. Increased risk of epidural/spinal hematoma secondary to systemic heparinization, potential hemodynamic instability, technical difficulties and complications such as pneumothorax are potential serious drawbacks. Due to the aforementioned reasons, anesthetists are understandably preferring ultrasound (US) guided interfascial plane blocks, which are generally thought to provide safer and more effective analgesia in cardiac surgery.

This study aims to evaluate and compare the effects of ESPB versus ESPB plus Superficial PIPB on pain scores and opioid consumption in patients undergoing elective cardiac surgery.

Patients will be divided into two groups:

Group ESPB:

In this group, patients will be administered bilateral ESPB (total of 40 ml, %0.25 bupivacaine) in addition to IV morphine patient-controlled analgesia (PCA) for the first 24 postoperative hours.

Group ESPB+Superficial PIPB:

In this group, patients will be administered Bilateral ESPB (total of 40 ml, %0.25 bupivacaine) and bilateral Superficial PIPB (total of 20 ml, %0.25 bupivacaine). In addition, IV morphine PCA will be administered for the first 24 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 2-3 patients between the ages of 18-80 who are scheduled for elective cardiac surgery (coronary artery bypass graft surgery +/- valve replacement or isolated valve surgery)
* BMI <35 kg / m2

Exclusion Criteria:

* Emergent surgeries, redo cases, minimally invasive procedures
* Patients who do not want to participate
* Patients with cognitive dysfunction (patients who are not able to evaluate the verbal numerical pain scale)
* Hypersensitivity or history of allergies to local anesthetics
* Major liver or kidney dysfunction or other pre-existing major organ dysfunction
* Left ventricular ejection fraction <30
* Individuals with mental health disorders (for example bipolar disorder or depression)
* Pregnancy or breastfeeding
* Presence of hematological disease
* Patients with alcohol-drug addiction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured. Patients will be able to request opioids via a PCA device when their NRS score ≥4.

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative day 1
  Pain at rest and while coughing will be assessed by numerical rating scale (NRS) scores at 0, 3, 6, 12, 18, and 24 hours after extubation. The NRS is an 11-point numeric scale that ranges from 0 to 10. The NRS is an 11-point scale consisting of integers from 0 to 10: 0 indicates "no pain" and 10 indicates "the worst pain ever possible." One day before the surgery, all patients will be informed about NRS and instructed on how to use a patient-controlled analgesia device.
Time to extubation | Postoperative day 1
  After the operation, the time until the patient is extubated will be recorded.
The number of patient requiring rescue analgesic | Postoperative Day 1
  The number of patients who required rescue analgesics will be recorded at 0, 3, 6, 12, 18, and 24 hours after extubation.
The incidences of post-operative nausea and vomiting (PONV) | Postoperative Day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more ondansetron 4 mg IV will be administered and will repeat after 8 hours if required.The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
Patient satisfaction as measured by the Revised American Pain Society Patient Outcome Questionnaire | Postoperative Day 1
  The Revised American Pain Society Patient Outcome Questionnaire will be used to assess satisfaction with pain expectation counseling (APS-POQ-R). The APS-POQ-R is designed for use in adult hospital pain management quality improvement activities, and it assesses six aspects of care: (1) pain severity and relief; (2) impact of pain on activity, sleep, and negative emotions; (3) side effects of treatment; (4) usefulness of pain treatment information; (5) ability to participate in pain treatment decisions; and (6) use of nonpharmacological strategies.
  Participants will rate themselves on a scale of 0 to 10. They were either severely dissatisfied or extremely satisfied, with a score of 0 indicating extreme dissatisfaction and 10 indicating extreme satisfaction.
  APS-POQ-R Turkish Version will be used for assessment.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients have any complications -directly related to the block or the drug used in the block- will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: BURHAN DOST, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Khera T, Murugappan KR, Leibowitz A, Bareli N, Shankar P, Gilleland S, Wilson K, Oren-Grinberg A, Novack V, Venkatachalam S, Rangasamy V, Subramaniam B. Ultrasound-Guided Pecto-Intercostal Fascial Block for Postoperative Pain Management in Cardiac Surgery: A Prospective, Randomized, Placebo-Controlled Trial. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):896-903. doi: 10.1053/j.jvca.2020.07.058. Epub 2020 Jul 24. PMID 32798172
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Derived] Dost B, Kaya C, Turunc E, Dokmeci H, Yucel SM, Karakaya D. Erector spinae plane block versus its combination with superficial parasternal intercostal plane block for postoperative pain after cardiac surgery: a prospective, randomized, double-blind study. BMC Anesthesiol. 2022 Sep 16;22(1):295. doi: 10.1186/s12871-022-01832-0. PMID 36114466